CLINICAL TRIAL: NCT00004030
Title: A Phase I/II Study of the Pharmacokinetics, Tolerability and Safety of Administration of VX-853 to Patients Receiving Single Agent Therapy With Doxorubicin HCI
Brief Title: VX-853 in Treating Patients With Solid Tumors Who Are Receiving Liposomal Doxorubicin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Marshall, MD, Georgetown University Medical Center
Purpose: Treatment
Other Study IDs: CDR0000065641; P30CA051008 (NIH); GUMC-96007; VX-95-853-001; VX-GUMC-96007; NCI-V97-1275
Record Dates: First submitted 1999-12-10; First posted 2004-05-25 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2001-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — timcodar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: VX-853
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of VX-853 in treating patients who have solid tumors who are receiving liposomal doxorubicin.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of VX-853 in combination with doxorubicin HCl liposome in patients with relapsed or incurable solid tumors. II. Obtain pharmacokinetic profiles for various dosages of VX-853 administered in combination with doxorubicin HCl liposome. III. Achieve whole blood concentrations of VX-853 in the predicted therapeutically effective range and characterize the pharmacokinetics at these doses. IV. Document antitumor effects of VX-853 in combination with doxorubicin HCl liposome in these patients.

OUTLINE: This is a dose escalation study of VX-853. Patients receive VX-853 orally every 8 hours on days 1-3 and doxorubicin HCL liposome IV over approximately 15 minutes beginning 26 hours after starting VX-853. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of VX-853 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued for this study within approximately 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven relapsed or incurable solid tumors No primary or metastatic CNS disease

PATIENT CHARACTERISTICS: See General Eligibility Criteria

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior cytotoxic chemotherapy (6 weeks since prior mitomycin or nitrosourea) Prior doxorubicin HCl allowed (no extensive therapy) Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Prior surgery allowed Other: Recovered from toxic effects of prior therapy At least 4 weeks since prior investigational or approved clinical trial agents No concurrent cimetidine, phenothiazines, phenytoin, calcium channel blockers, or cyclosporine or other P-glycoprotein inhibitors --Patients Characteristics-- Age: 18 and over Performance Status: Karnofsky 70-100% Life Expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Hemoglobin at least 9.0 g/dL Platelet count at least 100,000/mm3 Hepatic: AST and/or ALT no greater than 2 times upper limit of normal Bilirubin normal Renal: Creatinine normal Creatinine clearance at least 60 mL/min Cardiovascular: No clinically significant EKG abnormalities No atrial or ventricular arrhythmias requiring medication No ischemic event within 6 months of study Cardiac ejection fraction at least 50% by MUGA scan Other: Not pregnant or nursing Fertile patients must use effective contraception No prior or concurrent seizure disorders No prior or concurrent clinically significant medical illness No known hypersensitivity to doxorubicin HCl or other study medications No other active malignancies except curatively treated carcinoma in situ of the cervix or basal cell skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1996-03; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Hawkins, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (1):
- Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia, United States